CLINICAL TRIAL: NCT04679610
Title: Surveillance of in Vitro Activity of Ceftolozane-tazobactam Against Contemporary Nosocomial Gram-negative Pathogens Isolated in Russia
Brief Title: In Vitro Activity of Ceftolozane-tazobactam Against Contemporary Nosocomial Gram "-" Pathogens Isolated in Russia
Status: Completed | Type: Observational
Sponsor: The Interregional Association for Clinical Microbiology and Antimicrobial Chemotherapy (IACMAC) (Other)
Responsible Party: Sponsor
Other Study IDs: IAC-TOL/TAZ-2017-2020
Record Dates: First submitted 2020-12-08; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Nosocomial Infection
Keywords: ceftolozane-tazobactam, antibiotics, gram "-" bacteria, ESBL
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Infections caused by resistant gram-negative bacteria are becoming increasingly prevalent and now constitute a serious threat to public health worldwide because they are difficult to treat and are associated with high morbidity and mortality rates. Among nosocomial infections, the most major threat represent infections caused by multidrug-resistant (MDR) and extensively drug-resistant (XDR) Gram-negative pathogens.

DETAILED DESCRIPTION:
Infections caused by resistant gram-negative bacteria are becoming increasingly prevalent and now constitute a serious threat to public health worldwide because they are difficult to treat and are associated with high morbidity and mortality rates. Among nosocomial infections, the most major threat represent infections caused by multidrug-resistant (MDR) and extensively drug-resistant (XDR) Gram-negative pathogens. The most problematic are the ESKAPE microorganisms, an acronym of the most frequently isolated MDR bacteria (Enterococcus faecium, Staphylococcus aureus, Klebsiella pneumoniae, Acinetobacter baumannii, Pseudomonas aeruginosa and Enterobacter spp).

Extended-spectrum β-lactamases (ESBLs) have emerged as a major source of antimicrobial resistance in gram-negative pathogens. Generally encoded by plasmid-borne genes, these enzymes confer resistance to penicillins, cephalosporins, and aztreonam. In addition, their presence in bacteria has been associated with resistance to other classes of nonpenicillin antibiotics, including fluoroquinolones, aminoglycosides, trimethoprim-sulfamethoxazole, and β-lactam/β-lactamase inhibitor combinations. Thus, ESBL-producing organisms often possess a multidrug resistance phenotype. Furthermore ESBL production has been associated with severe adverse clinical and economic outcomes, including increased mortality, increased length of stay, delay in the institution of effective therapy, decreased functional status on discharge, and increased cost of care.

The recent emergence and spread of infections caused by carbapenem-resistant Enterobacteriaceae (CRE) are concerning because carbapenems have represented a last line of defense against resistant strains of gram-negative pathogens [6]. The most clinically relevant carbapenemases in Enterobacteriaceae are the class D enzymes of the OXA-48 group, class A enzymes of the KPC type and the zinc-dependent class B metallo-β-lactamases (MβLs), represented mainly by the VIM, IMP, and NDM type.

Carbapenemase-producing Enterobacteria cause serious infections in debilitated and immunocompromised patients, in association with prolonged hospital stays and increased mortality rates, ranging from 24% to as high as 70%, depending on the study population [8,9]. Given the critical condition of these patients, treatment should be timely and rapidly efficacious. However, therapeutic options are obviously limited.

The environmental bacterium P. aeruginosa is one of the most important nosocomial pathogens, especially in intensive care units. Intrinsic and acquired antibiotic resistance makes P. aeruginosa one of the most difficult organisms to treat. The high intrinsic antibiotic resistance of P. aeruginosa is due to several mechanisms: a low outer membrane permeability, the production of an AmpC β-lactamase, and the presence of numerous genes coding for different multidrug resistance efflux pumps[10]. Loss of OprD is the most prevalent mechanism of resistance to carbapenems and is associated with resistance to imipenem and reduced susceptibility to meropenem [11].

In the United States, there has been a steady increase since 2000 in rates of extended-spectrum β-lactamase-producing Enterobacteriaceae, carbapenem-resistant Enterobacteriaceae, and multidrug-resistant strains of Pseudomonas aeruginosa and Acinetobacter baumannii, particularly among hospitalized patients with intraabdominal infections, urinary tract infections, ventilator-associated pneumonia, and bacteremia [12].

In Russia there are some key issues of antimicrobial resistance according to the national multicenter surveillance study on antimicrobial resistance of nosocomial pathogens, "MARATHON" (2011-2012). Data were collected in 25 hospitals of 18 cities of Russia (1700 isolates). Enterobacteriaceae isolates jointly comprised 33.7% of all bacterial nosocomial isolates. Production of ESBL was detected in 78.2% of all isolates [13]. Thus there is an extremely high frequency of resistance to 3rd gen. cephalosporins in all species of Enterobacteriaceae (> 80%) and especially K. Pneumoniae (> 90%), due mainly spread of ESBL (78%), which complicates the possibility of their use in the empirical treatment of nosocomial infections caused by Enterobacteriaceae [14].

The level of resistance to carbapenems among Enterobacteriaceae was: non-susceptibility to meropenem - 2.8%, to imipenem - 8.4%, to ertapenem - 14.0%, including conferred by carbapenemases - 3.7% of isolates OXA-48 (3.3%), NDM (0.4%) [13].

Despite the fact that the carbapenems are active against most (86-97%) of nosocomial Enterobacteriaceae strains, the proportion of isolates resistant to carbapenems is increasing rapidly [14].

In Russia P. aeruginosa is the most common nosocomial pathogen, comprising 20.2% of all bacterial nosocomial isolates. The high level of resistance P. aeruginosa to carbapenems and high level of MBL were detected: resistance to imipenem - 88.0%, to meropenem - 66.8%, including resistance conferred by VIM-type MBL in 28.3% of the isolates [15].

The above date shows the need to develop novel antimicrobials. In an era of increasing resistance to antimicrobials, ceftolozane-tazobactam provides clinicians with an additional treatment option for infections caused by multidrug-resistant Gram-negative organisms, including ESBL-Enterobacteriaceae and carbapenem-resistant P. aeruginosa[16]. In vitro, ceftolozane-tazobactam has been shown to be active against P. aeruginosa and demonstrates high activity against Enterobacteriaceae [17]. Ceftolozane-tazobactam demonstrated in vitro activity against Enterobacteriaceae in the presence of some ESBLs and other betalactamases of the TEM, SHV,CTX-M, and OXA groups.

This study will assess the activity of ceftolozane-tazobactam against contemporary clinical isolates of the family Enterobacteriaceae and P. aeruginosa, including those with resistance to extended-spectrum cephalosporins and carbapenems. It will also assess the prevalence of various ESBLs of TEM-, SHV-, CTX-M- and GES-types, as well as carbapenemases of class A (KPC, GEScarb.), class D (OXA-48-like) and class B (NDM, VIM, IMP) and will evaluate the in vitro activities of ceftolozane-tazobactam and other antimicrobials against nosocomial isolates with respect to their beta-lactamase content. The results of this study will help to advance the understanding of ceftolozane-tazobactam's role in Russian hospitals.

ELIGIBILITY:
Inclusion Criteria:

* consecutive, non-duplicate (one per patient/episode of infection), gram-negative clinical isolates collected from patients with intra-abdominal, urinary tract, lower respiratory tract, and bloodstream nosocomial infections

Exclusion Criteria:

* Non-Enterobacteriaceae isolates after reidentification

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with gram-negative clinical isolates collected from patients with intraabdominal, urinary tract, lower respiratory tract, and bloodstream nosocomial infections
Sampling Method: Non-Probability Sample
Enrollment: 700 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
To access ceftolozane-tazobactam activity against many multidrug-resistant isolates of P. aeruginosa, | 01.01.2017 - 31.10.2018
  ceftolozane-tazobactam will demonstrate activity against many multidrug-resistant isolates of P. aeruginosa, including cephalosporin- and carbapenem-resistant isolates that do not produce a metallo-beta-lactamase
To access ceftolozane-tazobactam activity against P. aeruginosa producing class A ESBL | 01.01.2017 - 31.10.2018
  ceftolozane-tazobactam will demonstrate activity against P. aeruginosa isolates producing class A extended-spectrum beta-lactamases (ESBLs) and carbapenemases of GES type
To access ceftolozane-tazobactam activity against P. aeruginosa | 01.01.2017 - 31.10.2018
  ceftolozane-tazobactam will demonstrate activity against P. aeruginosa isolates of various genotypes including members of international high-risk clones
To determine the prevalence of Enterobacteriaceae producing extended-spectrum beta-lactamases (ESBLs) of molecular class A | 01.01.2017 - 31.10.2018
  the prevalence of Enterobacteriaceae producing extended-spectrum beta-lactamases (ESBLs) of molecular class A will be high
To determine the molecular class D (OXA-48-like) enzymes carbapenemases in Enterobacteriaceae in Russia and the prevalence of carbapenemases of molecular classes A and B | 01.01.2017 - 31.10.2018
  molecular class D (OXA-48-like) enzymes will be the most common carbapenemases in Enterobacteriaceae in Russia and the prevalence of carbapenemases of molecular classes A and B will be limited
To access ceftolozane-tazobactam activity against many Eterobacteriaceae isolates produsing ESBLs and/or OXA-48-like enzymes | 01.01.2017 - 31.10.2018
  ceftolozane-tazobactam will demonstrate activity againt many Eterobacteriaceae isolates produsing ESBLs and/or OXA-48-like enzymes

CONTACTS AND LOCATIONS:
Locations (1):
- The Interregional Association for Clinical Microbiology and Antimicrobial Chemotherapy, Smolensk, Russia